CLINICAL TRIAL: NCT07342543
Title: Guided Physical Activity Counseling for Hypertension in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Britta Larsen, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 811759
Record Dates: First submitted 2026-01-12; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Physical Activity; Hypertension; Prehypertension; Hypertension Grade I, Subgroup "Borderline" (WHO)
Keywords: primary care; physical activity counseling; fitness tracker; physical activity; prehypertension; stage 1 hypertension
MeSH Terms: conditions — Motor Activity; Hypertension; Prehypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Activity Counseling Guide (Experimental): Providers randomized to this group will provide physical activity counseling to patients based on their wearable fitness tracker data. Counseling will be guided by an online tool that synthesizes the patient's unique data and provides effective counseling prompts based on the data.
  Interventions: Behavioral: Physical activity counseling
- Standard of care (No Intervention): Providers randomized to this group will provide patients with the standard of care for physical activity counseling.
- Comparison: Fitbit Data Only (No Intervention): Providers randomly assigned to this group will have access to patients' Fitbit data but will not be provided with activity counseling prompts.

INTERVENTIONS:
Behavioral: Physical activity counseling — The personalized data system will use physical activity data from Fitbits to create summary system reports that will guide brief discussions between providers and patients regarding PA during clinic visits. To facilitate discussion, tailored guides for providers randomly assigned to the Intervention Arm will include each of the following elements: a) a visual summary of mean weekly minutes of MVPA over the past 4-6 weeks, b) whether they are meeting clinical guidelines of 150 minutes/week, c) whether their minutes are increasing, decreasing, or generally remaining the same, d) a script for performance feedback, e) questions tailored to whether the patient is increasing or decreasing their activity, f) a script to discuss an appropriate BCT through the lens of shared decision making, and g) a prompt to review the plan. The plan summary will be incorporated in the patient's after visit summary.
  Arms: Physical Activity Counseling Guide

SUMMARY:
The goal of this study is to create easy-to-read physical activity reports and counseling guides for primary care doctors. These tools will use activity data collected over time from wearable fitness trackers. The study will also test how helpful and easy the system is for doctors when talking with patients who have high blood pressure. This approach uses technology that already exists and helps solve problems that make it hard to use in medical care. It also has the potential to reach many people and be low-cost for clinics to use.

DETAILED DESCRIPTION:
There is robust evidence that adopting regular moderate-to-vigorous physical activity (MVPA) can improve blood pressure and reduce CVD risk in patients with hypertension. Accordingly, MVPA counseling is considered first line treatment for patients with pre- and stage 1 hypertension, though rates of counseling in ambulatory care visits for hypertension management remain low. Some health systems have begun incorporating data from wearable activity trackers (e.g., Fitbits) into electronic health records (EHR) to facilitate MVPA counseling, but it is unclear whether sharing these data with providers will change ambulatory care visits or patient behavior. Clinicians have reported myriad barriers to incorporating this technology into clinical care, including that reviewing data takes too much time, is not standardized, takes expertise they do not have, and there is often too much data to be useful. In addition to summarized data, providers may need guidance in how to interpret it, use evidence-based counseling practices, and suggest behavior change strategies based on patients' unique barriers. In the current proposal, investigators will conduct a 3-arm randomized trial to test the efficacy of an expert software system to interpret data from wearables for providers and generate tailored counseling scripts for them incorporating evidence-based communication strategies for primary care. The study team will recruit N=30 primary care providers from UC San Diego primary care clinics and N=300 of their patients with pre- and stage 1 hypertension (PS1H). All patients will receive a wearable Fitbit activity tracker to wear in the 4-6 weeks preceding an ambulatory care visit for PS1H management. Providers will be randomized to receive 1) algorithm-driven counseling guides in EHR with summarize data and tailored counseling scripts based on patient activity levels and barriers (intervention), 2) only summarized data from wearables integrated into EHR (comparison), or 3) no access to patient Fitbit data (control). Patients will continue to wear trackers continuously for 3 months following their ambulatory care visit, and will take at-home blood pressure readings monthly. Investigators hypothesize that patients whose providers are randomized to receive the expert system summary reports will show greater increases in MVPA following ambulatory care visits than those whose providers receive only summarized data and patients in the control group. The study team will also evaluate effects of the counseling guides on blood pressure, doctor-patient communication, and clinical workflow by using time stamps in EHR to estimate visit length. Investigators will also evaluate provider satisfaction with the system through questionnaires and interviews. This study will advance intervention science by creating an intervention tool for providers that has potential for low-cost implementation across a wide range of clinical settings. This will capitalize on the rich data that are increasingly generated by consumer wearables in clinical populations while addressing critical barriers to incorporating this data into clinical care.

ELIGIBILITY:
Inclusion Criteria for Providers:

1. Currently work for UC San Diego Health, with a primary appointment in one of the eight primary care clinics
2. Conduct ambulatory care visits for blood pressure management with at least 20 patients with a diagnosis of pre- or stage 1 hypertension

Inclusion Criteria for Patients:

1. Have received a diagnosis of pre- or stage 1 hypertension, and/or having SBP 120-139, DBP <89
2. be receiving care from one of the enrolled providers
3. be currently engaging in <150 minutes/week of at least moderate intensity exercise (see below)
4. be between age 18 and 80 years
5. not currently taking anti-hypertensive medication
6. able to read, speak, and understand English.

Exclusion Criteria for Providers:

1. planning to leave UCSD Health in the next 18 months
2. participated in the co-design workshops to design the PACE system
3. being unwilling to be randomized to one of the three conditions.

Exclusion Criteria for Patients:

1. any condition that would contraindicate unsupervised exercise as determined by their provider, such as severe cardiovascular or pulmonary disease limiting exercise tolerance
2. plans to change healthcare providers within the next two months
3. planned surgery or procedure that could impact mobility within the next five months
4. pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity Minutes Measured by Fitbit | 4 months
  Change in physical activity minutes measured by wrist-worn Fitbits in patients who that are assigned to providers receiving the PACE Guides during ambulatory care visits (intervention group) compared to those seeing providers in the comparison or control groups.

SECONDARY OUTCOMES:
Height in centimeters | Recorded at ambulatory care visit (4-6 weeks post-enrollment)
  Height in cm
Medication Use | 4 months
  Use and dose of medications per medical record
Blood Pressure (at-home) | 4 months
  Patients will be sent an Omron M10-IT blood pressure cuff for monthly at-home readings. They will be provided with detailed instructions and a link to an AHA video demonstrating proper measurement. Participants will measure BP twice, one minute apart, in a seated position after 5 minutes of rest. They will be instructed to measure at the same time of day each month, and to avoid caffeine or physical activity immediately before measurement. Readings will be shared via Bluetooth and recorded in a log.
Demographics (Patient) | Enrollment
  Age, race, ethnicity, education, income, marital status
Rate Your Plate | 4 months
  a 24-item tool capturing information regarding fat intake, animal and dairy protein, fruit, vegetables, whole grains, snacks, and sweets.
Social Support for Exercise (SSE) | 4 months
  Questionnaire measuring social support specifically in relation to exercise with three subscales (friends, family, rewards/punishments)
Self-Efficacy for Physical Activity (SE) | 4 months
  Questionnaire measuring confidence to become physically active across diverse contexts
Center for Epidemiologic Studies Depression Scale (CES-D) | 4 months
  20-item self reported questionnaire designed to measure depressive symptoms, with higher scores indicating possible depression
Perceived Stress Scale (PSS) | 4 months
  A 10-item scale used to assess stress levels with higher scores indicating greater perceived stress
Pittsburgh Sleep Quality Index | 4 months
  Questionnaire used to measure sleep quality
After-visit Questionnaire | immediately following ambulatory care visit in clinic (4-6 weeks post-enrollment)
  Assesses which topics were discussed during provider visit, including physical activity, goals, behavior change techniques, wearable tracker data, etc.
Communication and Shared Decision Making | immediately following ambulatory care visit in clinic (4-6 weeks post enrollment)
  the CollaboRATE questionnaire measuring patient experience of care, plus the facilitation subscale of the Perceived Involvement in Care scale
Fitbit Adherence | 4 months
  % of days Fitbit worn, % of days Fitbit synced within 5 days
Clinical Workflow | 2 months
  Timestamped user access logs in Epic to approximate visit lengths to assess if using the physical activity counseling guides impacts total visit timed
Consumer Satisfaction Questionnaire (Provider) | 18-36 months post-enrollment
  Assess overall satisfaction/acceptability and suggestions for improvement (intervention arm only)
Follow-up Interview (Provider) | 18-36 months post-enrollment
  A brief 20-minute interview to share experiences with the physical activity counseling guides (intervention arm) or summarized wearable data (comparison arm), and give suggestions for increased efficacy and usability
Demographics (Provider) | At enrollment
  Age, sex, provider type/degree, specialty, years in clinical practice
Weight in kg | Recorded at ambulatory care visit (4-6 weeks post-enrollment)
  Weight measured in kilograms
Resting blood pressure in clinic | Recorded at ambulatory care visit (4-6 weeks post-enrollment)
  Blood pressure in mm Hg as measured in clinic
Medication adherence | 4 months
  Medication Adherence Report Scale (MARS-5) is a 5-item questionnaire to assess self-reported adherence to medical regimens with higher scores indicating better adherence

IPD SHARING:
Plan to Share IPD: Yes
All quantitative data produced in the course of the project will be preserved and shared. Transcripts from stakeholder interviews will be shared only in the event that they give permission for the entire transcript to be shared; otherwise, summaries and codebooks will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 7 years after the end of the funding period.
Access Criteria: The Larsen USCD data provides metadata, persistent identifiers and long-term access. This repository is supported by USCD and dataset(s) are available through a request process directly with the PI, Dr. Larsen.